CLINICAL TRIAL: NCT00640510
Title: A Placebo-Controlled, Double-Blind Confirmatory Study of Rapid-Acting Intramuscular Olanzapine in Agitated Patients With Schizophrenia
Brief Title: A Study Comparing Rapid Acting Intramuscular Olanzapine and Placebo in Agitated Patients With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 9622; F1D-JE-RA03
Record Dates: First submitted 2008-03-18; First posted 2008-03-21 (Estimated); Results first posted 2009-08-26 (Estimated); Last update posted 2009-09-02 (Estimated); Status verified 2009-08

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Olanzapine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IM olanzapine 10mg (Experimental): Patients will receive at least one injection of Intramuscular (IM) olanzapine 10mg. If patients do not respond to the study medication or if patients do not have enough improvement based on the investigator's judgment, and in addition, if the investigator judges it is reasonable, the patient will receive a second injection at the same dose strength as the first injection after 2 hours following the first injection (no later than 8 hours after the first injection).
  Interventions: Drug: Rapid Acting Intramuscular Olanzapine
- IM placebo (Placebo Comparator): Patients will receive at least one injection of Intramuscular placebo. If patients do not respond to the study medication or if patients do not have enough improvement based on the investigator's judgment, and in addition, if the investigator judges it is reasonable, the patient will receive a second injection at the same dose strength as the first injection after 2 hours following the first injection (no later than 8 hours after the first injection).
  Interventions: Drug: Isotonic sodium chloride solution

INTERVENTIONS:
Drug: Rapid Acting Intramuscular Olanzapine — 10mg/injection, IM. If patients do not respond to the first study medication or if patients do not have enough improvement based on the investigator's judgment, and in addition, if the investigator judges it is reasonable, the patient will receive a second injection at the same dose strength as the first injection after 2 hours following the first injection (no later than 8 hours after the first injection).
  Other Names: LY170053; olanzapine; RAIM
  Arms: IM olanzapine 10mg
Drug: Isotonic sodium chloride solution — 0.9% sodium chloride (NaCl) solution. If patients do not respond to the first study medication or if patients do not have enough improvement based on the investigator's judgment, and in addition, if the investigator judges it is reasonable, the patient will receive a second injection at the same dose strength as the first injection after 2 hours following the first injection (no later than 8 hours after the first injection).
  Arms: IM placebo

SUMMARY:
The primary objectives of the study is to confirm if the efficacy of IM olanzapine in patients with schizophrenia is greater than IM placebo by comparing changes from baseline to 2 hours post first IM injection of agitation.

ELIGIBILITY:
Inclusion Criteria:

* Patients have met Diagnostic and Statistical Manual of Mental Disorders Fourth Edition, Text Revision (DSM-IV-TR) criteria for schizophrenia.
* Male or female, at least 20 years and less than 65 years old.
* Inpatients during the study.
* Each patient, or a proxy consenter, understand the nature of the study and must sign an informed consent document. The patient is able to cooperate with all study procedures in the view of the investigator.
* Patients are considered, by the investigator or subinvestigator, to be clinically agitated and appropriate candidates for treatment with intramuscular (IM) medication. The investigator must believe that it is safe to administer IM olanzapine to the patients with respect to the safety profile, including the anticholinergic properties of Olanzapine IM.
* Patients have a minimum total score of ≧ 20 on the five items of the Positive and Negative Syndrome Scale-Excited Component (PANSS-EC) using the 1-7 scoring system prior to the first injection of study drug.
* Patients have a score of 1 or 2 on the Agitation-Calmness Evaluation Scale (ACES) prior to the first injection of study drug.

Exclusion Criteria:

* Patients who were previously treated with oral olanzapine and are considered to be treatment-resistant to oral olanzapine, in the opinion of the investigator.
* Patients who have a history of allergic reaction or intolerance to study medication.
* Patients who show evidence of clinically significant bradycardia or arrhythmia obtained either from a physical exam or an electrocardiogram (ECG).
* Patients who require concomitant treatment with any other medication with primary central nervous system activity, other than those allowed as specified in section "concomitant treatment".
* Patients who have acute, serious or unstable medical conditions, including (but not limited to) hepatic insufficiency (specifically any degree of jaundice), recent cerebrovascular accidents, uncontrolled seizure disorders, serious acute systemic infection or immunologic disease, unstable cardiovascular disorders (including ischemic heart disease), renal, gastroenterologic, respiratory, endocrinologic, neurologic, or hematologic diseases.
* Patients with inadequately controlled diabetes, or patients whose treatment for diabetes were changed within 4 weeks prior to the first injection of the study drug. The investigator's discretion will supersede even if the patients do not meet the above criteria for concurrent diabetes.
* Patients who have a known neutrophil count or total of segmented cell and band cell counts of <1,500 /millimeter cubed (mm3).
* Patients who have a known alanine aminotransferase/serum glutamic pyruvic transaminase (ALT/SGPT) values ≧2 times the normal upper limit of the performing laboratory (ULN) or aspartate aminotransferase/serum glutamic oxaloacetic transaminase (AST/SGOT) values ≧3 times the ULN or total bilirubin values ≧1.5 times the ULN.
* Patients who have a known serum triglycerides ≧500 milligrams/deciliter (mg/dL).
* Electrocardiogram abnormalities considered clinically significant by the investigator.
* Patients who have had treatment with injectable depot antipsychotics within one injection interval prior to study drug administration.
* Patients who have received treatment with antipsychotics or other prohibited concomitant medicines showing in the section "prohibited concomitant medicines" within 2 hours prior to the first IM study drug administration.
* Patients who have had treatment with benzodiazepines within 4 hours prior to first IM study drug administration.
* Patients who have been administered epinephrine within 24 hours prior to the first IM study drug administration.
* Patients who have received treatment with psychostimulants or reserpine within 7 days prior to the first IM study drug administration.
* Patients who have received beta blockers or calcium channel blockers previously, must have been taking the same medication at the same dose for 28 days prior to the first IM study drug administration. No beta blockers or calcium channel blockers may be administered within 24 hours of the first IM study drug injection, or any time during the double blind phase.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2008-03; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (11):
- Japan (11):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukushima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gunma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kagoshima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kumamoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Okayama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Okinawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saga
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tottori
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yamagata

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One patient randomized to placebo was withdrawn from study by physician and is not included in the baseline demographic data table.
Groups:
- IM Olanzapine 10mg: Patients will receive at least one injection of Intramuscular olanzapine 10mg. If patients do not respond to the study medication or if patients do not have enough improvement based on the investigator's judgment, and in addition, if the investigator judges it is reasonable, the patient will receive a second injection at the same dose strength as the first injection after 2 hours following the first injection (no later than 8 hours after the first injection).
Period: Overall Study
Arm/Group | IM Olanzapine 10mg | IM Placebo
Started | 17 | 17 (One patient randomized to placebo discontinued prior to receiving study drug.)
Completed | 16 | 15
Not Completed | 1 | 2
Not completed — Lack of Efficacy | 0 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IM Olanzapine 10mg | IM Placebo | Total
Number analyzed (Participants) | 17 | 16 | 33
Age Continuous [Mean (Standard Deviation); unit: years] | 47.4 (12.4) | 45.9 (11.5) | 46.7 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 9 | 10 | 19
Region of Enrollment [Number; unit: participants]
  Japan | 17 | 16 | 33
Diabetes Mellitus [Number; unit: participants]
  Yes | 2 | 2 | 4
  No | 15 | 14 | 29
Diagnostic and Statistical Manual of Mental Disorders Fourth Edition, Text Revision Diagnosis [Number; unit: participants]
  Catatonic | 2 | 0 | 2
  Disorganized | 7 | 7 | 14
  Paranoid | 7 | 7 | 14
  Undifferentiated | 1 | 0 | 1
  Residual | 0 | 2 | 2
Pre-Therapy Antipsychotic Usage [Number; unit: participants]
  Yes (>=1000 milligrams/day) | 7 | 6 | 13
  Yes (<1000 milligrams/day) | 9 | 9 | 18
  No | 1 | 1 | 2
Age at Onset [Mean (Standard Deviation); unit: years] | 22.6 (6.4) | 21.3 (6.1) | 22.0 (6.2)
Agitation-Calmness Evaluation Scale (ACES) [Mean (Standard Deviation); unit: units on a scale] — The ACES differentiates agitation, calmness, and sleep-state, using a 9-point scale: 1 (Marked Agitation) to 9 (Unarousable).
  units on a scale | 1.8 (0.4) | 1.8 (0.4) | 1.8 (0.4)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms/square centimeters] — Body mass index is an estimate of body fat based on body weight divided by height squared.
  kilograms/square centimeters | 20.7 (2.9) | 22.8 (3.6) | 21.7 (3.3)
Positive and Negative Syndrome Scale-Excited Component [Mean (Standard Deviation); unit: units on a scale] — Measures excitability and consists of the following 5 items from the PANSS: Excitement, Hostility, Tension, Uncooperativeness, and Poor Impulse Control. Each item is rated on a scale from 1 (Absent) to 7 (Extreme). The sum of the 5 items is defined as the PANSS-EC total score which ranges from 5 to 35.
  units on a scale | 23.6 (3.8) | 23.5 (3.8) | 23.5 (3.7)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 2 Hours Post the First Intramuscular (IM) Injection in Positive and Negative Syndrome Scale-Excited Component (PANSS-EC)
Description: Measures excitability and consists of the following 5 items from the PANSS: Excitement, Hostility, Tension, Uncooperativeness, and Poor Impulse Control. Each item is rated on a scale from 1 (Absent) to 7 (Extreme). The sum of the 5 items is defined as the PANSS-EC total score which ranges from 5 to 35.
Time Frame: 2 hours post first intramuscular (IM) injection
Population: Number of randomized patients having the measures both at baseline and post-baseline. Last Observation Carried Forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IM Olanzapine 10mg | IM Placebo
Number analyzed (Participants) | 16 | 16
units on a scale | -4.7 (4.8) | -4.6 (4.5)
Statistical Analysis 1: Comparison: IM Olanzapine 10mg vs IM Placebo; A sample size of at least 15 patients per group was necessary to verify that the decrease in PANSS-EC total score was significantly greater in the IM olanzapine group than the placebo group using Student's t-test with a power of 90% at a two-sided significance level of 5%; Test type: Superiority or Other; p = 0.940, t-test, 2 sided

2. Secondary Outcome: Change From Baseline to Each Timepoint in Positive and Negative Syndrome Scale-Excited Component (PANSS-EC)
Description: as for outcome 1
Time Frame: 15 min, 30 min, 60 min, 90 min post first IM injection
Population: Number of patients having the measure both at baseline and post-baseline. Last Observation Carried Forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IM Olanzapine 10mg | IM Placebo
Number analyzed (Participants) | 16 | 16
units on a scale
  Change from Baseline to 15 minutes | -1.2 (1.3) | -1.2 (1.5)
  Change from Baseline to 30 minutes | -2.9 (2.8) | -2.4 (2.8)
  Change from Baseline to 60 minutes | -3.8 (3.6) | -3.4 (4.1)
  Change from Baseline to 90 minutes | -5.1 (4.3) | -4.6 (4.7)
Statistical Analysis 1: Comparison: IM Olanzapine 10mg vs IM Placebo; Test type: Superiority or Other; p = 1.000, t-test, 2 sided — P-value for Change from Baseline to 15 minutes. Change = Timepoint minus Baseline
Statistical Analysis 2: Comparison: IM Olanzapine 10mg vs IM Placebo; Test type: Superiority or Other; p = 0.620, t-test, 2 sided — P-value for Change from Baseline to 30 minutes. Change = Timepoint minus baseline
Statistical Analysis 3: Comparison: IM Olanzapine 10mg vs IM Placebo; Test type: Superiority or Other; p = 0.784, t-test, 2 sided — P-value for Change from Baseline to 60 minutes. Change = Timepoint minus baseline
Statistical Analysis 4: Comparison: IM Olanzapine 10mg vs IM Placebo; Test type: Superiority or Other; p = 0.756, t-test, 2 sided — P-value for Change from Baseline to 90 minutes. Change = Timepoint minus baseline

3. Secondary Outcome: Number of Responders at 2 Hours After First Intramuscular (IM) Injection
Description: A responder was defined ast he patient with ≥ 40% decrease in the PANSS-EC total score at 2 hours after the first IM injection in comparison with baseline. (See outcome measure 1 for description of PANSS-EC).
Time Frame: 2 hours post first IM injection
Population: Number of patients having the measures both at baseline and post-baseline. Last Observation Carried Forward.
Measure: Number; unit: participants
Arm/Group | IM Olanzapine 10mg | IM Placebo
Number analyzed (Participants) | 16 | 16
participants | 3 | 4
Statistical Analysis 1: Comparison: IM Olanzapine 10mg vs IM Placebo; Test type: Superiority or Other; p = 1.000, Fisher Exact

4. Secondary Outcome: Number of Participants With Scores of 4 to 7 in the Agitation-Calmness Evaluation Scale (ACES) at Each Timepoint
Description: The ACES differentiates agitation, calmness, and sleep-state, using a 9-point scale: 1 (Marked Agitation) to 9 (Unarousable). Scores of 4 (Normal) to 7 (Marked Calmness) were used for this outcome measure.
Time Frame: 30 min, 60 min, 90 min and 2 hours post first IM injection
Population: Number of patients having the measure at post-baseline. Last Observation Carried Forward.
Measure: Number; unit: participants
Arm/Group | IM Olanzapine 10mg | IM Placebo
Number analyzed (Participants) | 16 | 16
participants
  30 Minutes | 1 | 1
  60 Minutes | 1 | 1
  90 Minutes | 2 | 2
  2 Hours | 3 | 2
Statistical Analysis 1: Comparison: IM Olanzapine 10mg vs IM Placebo; Test type: Superiority or Other; p = 1.000, Fisher Exact — P-value for 30 Minutes
Statistical Analysis 2: Comparison: IM Olanzapine 10mg vs IM Placebo; Test type: Superiority or Other; p = 1.000, Fisher Exact — P-value for 60 Minutes
Statistical Analysis 3: Comparison: IM Olanzapine 10mg vs IM Placebo; Test type: Superiority or Other; p = 1.000, Fisher Exact — P-value for 90 Minutes
Statistical Analysis 4: Comparison: IM Olanzapine 10mg vs IM Placebo; Test type: Superiority or Other; p = 1.000, Fisher Exact — P-value for 2 Hours

ADVERSE EVENTS:
Arm/Group | IM Olanzapine 10mg | IM Placebo
Serious Adverse Events (participants affected / at risk) | 0 | 0
Other Adverse Events (participants affected / at risk) | 4 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | IM Olanzapine 10mg | IM Placebo
Blood creatine phosphokinase increased (Investigations) | 0/17 (0) | 1/16 (1)
Blood glucose increased (Investigations) | 1/17 (1) | 0/16 (0)
Blood pressure increased (Investigations) | 1/17 (1) | 0/16 (0)
Electrocardiogram T wave inversion (Investigations) | 0/17 (0) | 1/16 (1)
Glucose urine present (Investigations) | 1/17 (1) | 0/16 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1/17 (1) | 0/16 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days